CLINICAL TRIAL: NCT00722410
Title: Safety and Efficacy Study of Eradication of Carbapenem Resistant Klebsiella Pneumonia From the Gastrointestinal Tract by Probiotics.
Brief Title: Probiotics for Eradication of Carbapenem Resistant Klebsiella Pneumonia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Maya Margalit, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRKP-HMO-CTIL
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Anti-Biotic Resistance; Klebsiella Pneumoniae
Keywords: Carbapenem; resistant; Klebsiella pneumoniae; Carpapenemases; Probiotics; VSL3
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (No Intervention)
- B (Experimental): VSL#3 for 4 weeks
  Interventions: Dietary Supplement: VSL#3
- C (Experimental): Mechanical bowel cleansing followed by VSL#3 for 4 weeks.
  Interventions: Dietary Supplement: VSL#3; Drug: Polyethylene glycol

INTERVENTIONS:
Dietary Supplement: VSL#3 — A probiotic preparation.
  Arms: B; C
Drug: Polyethylene glycol — Oral ingestion of 3 liters of polyethylene glycol solution.
  Other Names: New Meroken.; Precolonoscopy solution.
  Arms: C

SUMMARY:
Infection by Klebsiella pneumonia producing class A carbapenemases is a major clinical and public health problem in Israel and worldwide. The aim of this study is to determine the safety and efficacy of alteration of the gut microflora by probiotics, alone or in combination with mechanical bowel cleansing, as a strategy to eradicate colonization of the gastrointestinal tract by CRKP. We hypothesize that administration of probiotics will decrease the rate of GI colonization by CRKP.

DETAILED DESCRIPTION:
CRKP colonization will be determined by culture and PCR of rectal swabs. The study will include 3 arms - no intervention, probiotics and mechanical bowel cleansing + probiotics. Followup examination of rectal swab samples for the presence of CRKP will be performed at 4 weeks and 12 weeks from study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are > 18 years of age.
2. Signing of informed consent by subject or legal custodian.
3. Colonization of the gastrointestinal tract by CRKP as determined by stool culture or PCR of stool for the blakpc gene.
4. Negative cultures for CRKP from extra-intestinal sites excluding urine.

Exclusion Criteria:

1. Subjects who have participated in another clinical trial within the last three months.
2. Women with childbearing potential unless using adequate contraception (IUD, oral or depot contraceptive or barrier plus spermicide).
3. Subjects who are pregnant or breast feeding.
4. Subjects who will be unavailable for the duration of the trial, are likely to be non-compliant with the protocol, or who are felt to be unsuitable by the investigator for any other reason.
5. Subjects with chronic diarrhea (>4 weeks).
6. Subjects with inflammatory bowel disease.
7. Subjects whose stool is positive for Clostridium difficile toxin.
8. Subjects receiving immunosuppressive treatment (i.e. corticosteroids; azathioprine or 6-MP; cyclosporine; tacrolimus; OKT3, methotrexate; anti TNF agents; chemotherapy).
9. Subjects who underwent solid organ or hematopoietic stem cell transplantation.
10. Subjects with primary or secondary immunodeficiency disorders, including HIV.
11. Subjects with chronic advanced cardiac, respiratory, renal or liver disease.
12. Subjects with advanced malignant disease.
13. Subjects with severe acute organ failure.
14. Subjects in whom CRKP is isolated from sites other than stool or urine (i.e. blood, sputum or wound cultures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
A negative stool culture for Carbapenem resistant Klebsiella pneumonia. | 4 weeks.

SECONDARY OUTCOMES:
A negative stool culture and/or PCR assay for CRKP at twelve weeks after initiation of probiotics (i.e - 8 weeks after cessation of probiotic treatment). | 12 weeks beginning of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Margalit, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Leavitt A, Navon-Venezia S, Chmelnitsky I, Schwaber MJ, Carmeli Y. Emergence of KPC-2 and KPC-3 in carbapenem-resistant Klebsiella pneumoniae strains in an Israeli hospital. Antimicrob Agents Chemother. 2007 Aug;51(8):3026-9. doi: 10.1128/AAC.00299-07. Epub 2007 Jun 11. PMID 17562800
- [Background] Manley KJ, Fraenkel MB, Mayall BC, Power DA. Probiotic treatment of vancomycin-resistant enterococci: a randomised controlled trial. Med J Aust. 2007 May 7;186(9):454-7. doi: 10.5694/j.1326-5377.2007.tb00995.x. PMID 17484706